CLINICAL TRIAL: NCT07003997
Title: Janus Kinase (JAK) Signaling in Depression
Brief Title: JAK Signaling in Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Felger, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009295; 1R01MH140180-01 (NIH)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — baricitinib; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baricitinib Arm (Experimental): Baricitinib at dose of 2 mg will be dispensed to be taken orally, daily for 8 weeks.
  Interventions: Drug: Baricitinib
- Placebo Arm (Placebo Comparator): Placebo will be dispensed to be taken orally, daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — This small molecule, orally bioavailable agent is an immunosuppressant (a medicine that reduces the activity of the immune system). It works by blocking the action of enzymes known as Janus kinases (JAK). These enzymes play an important role in the processes of inflammation. Patients will receive a dose of 2 mg oral daily.
  Other Names: Olumiant
  Arms: Baricitinib Arm
Drug: Placebo — A placebo is a sugar pill that has no therapeutic effect and will be administered orally. Participants will receive 1 placebo tablet matching the baricitinib tablet.
  Other Names: Sugar pill
  Arms: Placebo Arm

SUMMARY:
This study will test the hypothesis that Janus kinase (JAK) signaling is involved in major depression (MD) with high inflammation by determining whether its inhibition with baricitinib can improve functional connectivity in reward and motor circuits in association with improved motivation and motor function in MD patients enriched for high C-reactive protein (CRP) and anhedonia.

DETAILED DESCRIPTION:
Many people with depression also have high inflammation, which may be a cause of some of their depression symptoms. This study is being done to learn how inflammation affects the brain to cause symptoms of depression like anhedonia, low motivation and motor slowing. This will be tested using a medication called baricitinib that blocks one aspect of inflammation involving Janus kinase (JAK) signaling. The population to be included in this study are patients with depression and symptoms of anhedonia who have high inflammation as determined by a blood test. Patients must also be free of uncontrolled medical illnesses. Patients enrolled in the study will be randomly treated with either baricitinib or a placebo (matching sugar pill) for 8 weeks and assessed for markers of inflammation in the blood and symptoms of depression using self-reported and clinician-guided assessments. In addition, brain scans and computerized testing will be done to measure brain function and levels of motivation and motor speed. Participation in the study will include at least 8 visits over 2-3 months, including screening. Subjects will be recruited from local clinics and from the Atlanta community using social media ads. Approximately 100 subjects will be enrolled for this study to obtain 60 subjects who will be randomized to baricitinib or placebo. Blood and information from the brain scans, computerized testing and assessments of depression will be saved for future use. Consent to participate in the study will be obtained either remotely or in person by a trained staff member.

ELIGIBILITY:
Inclusion Criteria:

1. willing and able to give written informed consent;
2. men or women, 25-55 years of age;
3. a primary diagnosis of DSM-V major depression, current, or Bipolar, depressed type as diagnosed by the SCID-V;
4. score of >14 on the PHQ-9 from screening and HAM-D score ≥18 for study entry;
5. off all antidepressant or other psychotropic therapy (e.g. mood stabilizers, antipsychotics, and sedative hypnotics) for at least 4 weeks prior to baseline visit (8 weeks for fluoxetine),
6. CRP ≥3 mg/L,
7. PHQ-9 anhedonia score ≥2.

Exclusion Criteria:

1. history or evidence (clinical and laboratory) of an autoimmune disorder
2. history or evidence (clinical or laboratory) of hepatitis B or C infection or human immunodeficiency virus infection;
3. history of any type of cancer requiring treatment with more than minor surgery;
4. unstable cardiovascular, endocrinologic, hematologic, hepatic, renal, or neurologic disease (as determined by physical examination, EKG and laboratory testing);
5. significant hematological abnormalities at screening (ANC < 1500, Hgb<10, platelet< 100,000)
6. history of progressive multifocal leukoencephalopathy,
7. history of deep venous thrombosis,
8. history of cardiovascular disease (coronary artery disease, congestive heart failure, stroke - controlled hypertension is OK),
9. major surgery within 8 weeks prior to screening or will require major surgery during the study,
10. current or recent (<4 weeks prior to randomization) viral (including COVID-19), bacterial, fungal, or parasitic infection or any other active or recent infection,
11. symptomatic herpes zoster infection at or within 12 weeks of randomization,
12. history of disseminated/complicated herpes zoster (for example, ophthalmic zoster or CNS involvement),
13. cirrhosis of the liver from any cause,
14. any of the following specific abnormalities on screening laboratory tests: ALT or AST >2 x upper limits of normal (ULN), alkaline phosphatase (ALP) ≥2 x ULN, total bilirubin ≥1.5 x ULN (with the exception of patients on atazanavir, who must have total bilirubin <2 x ULN),
15. chronic kidney disease with eGFR <60 mL/min/1.73 m2,
16. history of any (non-mood-related) psychotic disorder; active psychotic symptoms of any type; substance abuse/dependence within 6 months of study entry (as determined by standardized clinician interview);
17. active suicidal plan as determined by a score >3 on item #3 on the HAM-D; g. an active eating disorder (except for patients with binge eating disorder in whom binging is clearly associated with worsening of mood symptoms);
18. history of a cognitive disorder or traumatic head injury involving loss of consciousness;
19. pregnancy or lactation,
20. use of gender affirming hormone therapy;
21. chronic use of non-steroidal anti-inflammatory agents (NSAIDS) (excluding 81mg of aspirin), immunosuppressive (e.g., biologics), glucocorticoid containing medications or minocycline within 6 months, or non-prescription supplements with known or suspected anti-inflammatory properties (e.g. fish oil supplements) within 2 weeks of baseline, or at any time during the study;
22. any contraindication for MRI scanning;
23. failure of more than 2 antidepressant trials (at least 6 weeks at recommended dose) in the current episode or 5 antidepressant trials lifetime; and
24. BMI >45 (to exclude severe obesity) or at the PI's discretion based on the patient's ability to fit comfortably in the MRI scanner.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Change in corticostriatal FC in reward and motor circuits after 2 and 8 weeks of study medication | Baseline, week 2 and 8 post-intervention
  FC in the corticostriatal circuits will be calculated as the degree of correlation in activity using a priori defined seeds in ventral and dorsal striatum and regions of interest (ROIs) in ventromedial prefrontal cortex (vmPFC) and pre-supplementary motor area (SMA). FC is measured as continuous Z scores reflecting the correlation of activity between the brain regions. Higher FC Z scores reflect stronger connectivity.

SECONDARY OUTCOMES:
Change in Effort Expenditure for Reward (EEfRT) | Baseline, 2, 4 and 8 weeks post-intervention
  The EEfRT is a widely used, multi-trial task measuring motivation for rewards as an assessment of anhedonia, as anhedonia is specifically associated with decreased motivation for rewards.
  Participants are given an opportunity to choose between two different task difficulty levels in order to obtain monetary rewards by repeated manual button presses within a short time. Button presses raises a virtual ''bar'' viewed onscreen. If they raise the bar to the ''top'' within the prescribed time, they are eligible to win the allotted money. Each trial presents the subject with a choice between two levels of task difficulty, a 'hard task' and an 'easy task' and 3 probabilities of winning. Subjects participate in the task for 20 minutes and the first 50 trials are analyzed by calculating proportion of hard-task choices across each level of probability. Lower proportions of hard task choices indicate decreased motivation.
Change in Finger Tapping Task (FTT) | Baseline, 2, 4 and 8 weeks post-intervention
  This task uses a specially adapted tapper that the subject is asked to tap as fast as possible using the index finger. The subject is given 5 consecutive 10-second trials for both the preferred and non-preferred hands. The finger tapping score is the mean of the 5 trials and is computed for each hand.
  A lower score indicates motor impairment.
Change in Trail Making Tests A (TMT) | Baseline, 2, 4, and 8 weeks post-intervention
  In Trail Making Test (TMT) Part A, the participant is tasked with drawing a continuous line connecting a series of 25 numbered circles in ascending order, from 1 to 25. This part of the test primarily assesses visual attention, processing speed, and visuomotor skills. Scoring is based on the time it takes to complete the task, measured in seconds. Higher scores reflect greater impairment or slower completion time (worse outcome).
Change in Inventory of Depressive Symptoms Self Report (IDS-SR) Anhedonia Subscale Score | Baseline, 2, 4, 6 and 8 weeks post-intervention
  Anhedonia is assessed with a 3-item subscale of the Inventory of Depressive Symptomatology Self-Report (IDS-SR). Items are scored on a 4-point scale from 0 to 3. Total scores for the Anhedonia Subscale range from 0 to 9 with higher scores reflecting greater anhedonia.
Change in Snaith-Hamilton Pleasure Scale-Clinician (SHAPS-C) score | Baseline, 2, 4, 6 and 8 weeks post-intervention
  SHAPS-C is a 14-item clinician-administered scale that assesses a patient's ability to experience pleasure, specifically in the context of anhedonia (loss of pleasure) and depression. Consists of 14 questions that the clinician asks the patient, with each question having a set of response categories (e.g., "Strongly Agree," "Agree," "Disagree," "Strongly Disagree"). Answers are scored based on whether the patient agrees or disagrees with the statement, with a score of 1 for disagreement (indicating a difficulty experiencing pleasure) and 0 for agreement. Total scores range from 0-14, with higher scores indicating greater difficulty experiencing pleasure or a higher level of anhedonia.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Felger, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier for the NIMH Data Archive (NDA) will also be collected for each subject.
Time Frame: The research community will have access to data at the end of the grant award or when a publication has been submitted. Once the data are submitted to NDA, that archive will control the long-term persistence of the data set. Currently, NDA has no process for deleting or retiring data sets.
Access Criteria: Data will be findable for the research community through the NDA Collection that will be established when this application is funded.
  To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.